CLINICAL TRIAL: NCT01781039
Title: Investigation of Anatomical Correlates of Speech Discrimination
Status: Recruiting | Type: Observational
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Responsible Party: Principal Investigator, Mark Parker, Director of Audiology, St. Elizabeth's Medical Center, Steward St. Elizabeth's Medical Center of Boston, Inc.
Other Study IDs: 00652
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Sensorineural Hearing Loss
Keywords: "hair cell"; "hearing aid"; "hearing loss"; "auditory nerve"; synaptopathy; "Outer hair cell"; "Otoacoustic emission"
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss; Vestibulocochlear Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- low HIN difficulty- anesthetized: Subjects with normal OHC function and who will be undergoing an previously scheduled anesthetized procedure will be assigned into 2 groups based on their self-perceived HIN difficulty (high and low difficulty), and then undergo a test battery consisting of auditory threshold tests, objective HIN assays, OHC measurements, cognitive processing, and central auditory processing evaluations. Immediately after anesthetization, electrocochleography (ECochG) will be used to measure CAP amplitudes, which will be correlated with measurements obtained from unanesthetized subjects as described below. This aim will determine the optimal CAP recording method with the strongest correlation with HIN performance in humans
- high HIN difficulty- anesthetized: Subjects with normal OHC function and who will be undergoing an previously scheduled anesthetized procedure will be assigned into 2 groups based on their self-perceived HIN difficulty (high and low difficulty), and then undergo a test battery consisting of auditory threshold tests, objective HIN assays, OHC measurements, cognitive processing, and central auditory processing evaluations. Immediately after anesthetization, electrocochleography (ECochG) will be used to measure CAP amplitudes, which will be correlated with measurements obtained from unanesthetized subjects as described below. This aim will determine the optimal CAP recording method with the strongest correlation with HIN performance in humans
- Hearing Aid fitting: MAD: Microphone adaptive directionality (MAD) feature will be activated, the WDC set to linear, and the DNR minimized
  Interventions: Device: Hearing Aid fitting
- Hearing Aid fitting: WDC: Wide dynamic compression (WDC) feature will be set to target levels, the MAD feature set to omnidirectional, and the DNR minimized.
  Interventions: Device: Hearing Aid fitting
- Hearing Aid fitting: DNR: Digital noise reduction (DNR) set to maximum, MAD set to omnidirectional, and WDC set to linear
  Interventions: Device: Hearing Aid fitting
- Hearing Aid fitting: Positive control: All hearing aid features enables
  Interventions: Device: Hearing Aid fitting
- Hearing Aid fitting: Negative control: All hearing aid features disabled
  Interventions: Device: Hearing Aid fitting

INTERVENTIONS:
Device: Hearing Aid fitting — Subjects with hfPTAs ranging from 0-55 dB HL will be recruitedwith 100 persons self-reporting difficulty HIN (> 50% of the time), and 100 persons reporting little difficulty HIN (< 50% of the time) will be randomly assigned to one of five groups (n = 200) based on enabled HA features using an online random assignment tool. Unaided HIQ and HIN assessments will be conducted in the sound field, and baseline DPOAE and CAP assessments will be measured. Subjects will be fit with binaural premium level receiver-in-the canal HAs (Phonak B90 or equivalent model at the start of the study) with 56 dB SPL gain receivers, using closed domes, and programmed to NAL-NL2 target gain, and randomly assigned to the groups.
  Groups: Hearing Aid fitting: DNR; Hearing Aid fitting: MAD; Hearing Aid fitting: Negative control; Hearing Aid fitting: Positive control; Hearing Aid fitting: WDC

SUMMARY:
Understanding speech is essential for good communication. Individuals with hearing loss and poor speech discrimination often have little success with hearing aids because amplifying sound improves audibility, but not clarity of the speech signal. The purpose of this study is to determine the relative importance of the sensory cells of the inner ear and auditory neurons on speech discrimination performance in quiet and in noise. This information may be used as a predictor of hearing aid benefit. The investigators expect to find decreased speech understanding ability resulting from both loss of sensory cells and the loss of auditory neurons.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing to moderate sensorineural hearing loss
* Sufficient English proficiency to complete speech discrimination testing in English

Exclusion Criteria:

* Hearing loss less than a 45 dB HL pure tone average (average hearing thresholds at 500, 1000 and 2000 Hz)
* Conductive hearing loss
* Neurodegenerative disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients referred from the St. Elizabeth's Department of Otolaryngology and self-referred patients to the Audiology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 1652 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Regression analysis | June 2024
  Regression analysis will be used to look for a correlation between measures of sensory cell and auditory neuron survival and speech recognition performance.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Parker, PhD, Principal Investigator — Steward St. Elizabeth's Medical Center
Locations (1):
- Steward St. Elizabeth's Medical Center, Brighton, Massachusetts, United States

REFERENCES:
- [Result] Bramhall N, Ong B, Ko J, Parker M. Speech Perception Ability in Noise is Correlated with Auditory Brainstem Response Wave I Amplitude. J Am Acad Audiol. 2015 May;26(5):509-517. doi: 10.3766/jaaa.14100. PMID 26055840
- [Result] Hoben R, Easow G, Pevzner S, Parker MA. Outer Hair Cell and Auditory Nerve Function in Speech Recognition in Quiet and in Background Noise. Front Neurosci. 2017 Apr 7;11:157. doi: 10.3389/fnins.2017.00157. eCollection 2017. PMID 28439223
- [Result] Parker MA. Identifying three otopathologies in humans. Hear Res. 2020 Dec;398:108079. doi: 10.1016/j.heares.2020.108079. Epub 2020 Sep 24. PMID 33011456
- See also: Peer reviewed publication — http://dx.doi.org/10.3766/jaaa.14100
- See also: Peer reviewed publication — https://www.frontiersin.org/articles/10.3389/fnins.2017.00157/full
- See also: Peer reviewed publication — https://doi.org/10.1016/j.heares.2020.108079

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT01781039/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT01781039/SAP_001.pdf